CLINICAL TRIAL: NCT00333385
Title: Continuous Versus Short Infusions of Ceftazidime in Cystic Fibrosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche (Other)
Collaborators: Vaincre la Mucoviscidose (Other); GlaxoSmithKline (Industry); Baxter Healthcare Corporation (Industry); Roche Pharma AG (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 01648
Record Dates: First submitted 2006-06-02; First posted 2006-06-05 (Estimated); Last update posted 2006-06-05 (Estimated); Status verified 2001-03

CONDITIONS: Cystic Fibrosis; Pseudomonas Aeruginosa; Pulmonary Exacerbation
Keywords: Ceftazidime; Continuous infusion; Antibiotic course
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections | interventions — Ceftazidime

INTERVENTIONS:
Drug: ceftazidime

SUMMARY:
The aim of this trial was to compare the safety and efficacy of courses of tobramycin and ceftazidime, administered intravenously as either thrice daily short infusions or 24 h continuous infusion, in cystic fibrosis patients with acute exacerbation of chronic pulmonary PA infection. In conventional treatment regimens, ceftazidime is administered in the form of thrice daily short infusions, but pharmacodynamic considerations suggest that continuous infusion could be more effective.

DETAILED DESCRIPTION:
Each patient received two successive IV antibiotic courses during a period of pulmonary exacerbation. One of these courses was delivered as thrice daily 30-minute infusions of ceftazidime in 100 ml of 0.9% sodium chloride, and the other was delivered as a continuous infusion of ceftazidime in 230 ml of 0.9% sodium chloride, over 23 hours. The daily dose of ceftazidime was 200 mg/kg, with a maximum dose of 12 g. For ceftazidime continuous infusion, a loading dose of 60 mg/kg (maximum 2 g) was used. All patients also received tobramycin (10 mg/kg), in the form of one 30-minute infusion per day. Portable devices were used: Intermate® SV 200 (Baxter) for the 30-minute short infusions of ceftazidime and tobramycin, Infusor® LV10 (Baxter) for continuous infusion of ceftazidime.

ELIGIBILITY:
Inclusion Criteria:

* patients with cystic fibrosis older than 8 years
* with chronic Pseudomonas aeruginosa infection of the respiratory tract
* with at least 2 courses of IV antibiotic in the year before enrolment
* at the time of a pulmonary exacerbation

Exclusion Criteria:

* allergy to ceftazidime or tobramycin
* bronchial colonization with Burkholderia cepacia
* renal impairment
* history of lung transplantation

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2001-10; Study Completion 2004-04

PRIMARY OUTCOMES:
Change in forced expiratory volume in 1s (FEV1) between the beginning and the end of the IV antibiotic course, expressed as a percentage of the predicted normal value

SECONDARY OUTCOMES:
the interval between 2 successive IV antibiotic courses
quality of life scores
sputum collected at the beginning and the end of each antibiotic course
plasma ceftazidime concentration at steady state (Css) for ceftazidime continuous infusion, and before (C trough), 30 minutes (Cmax) and 4 hours after (C4) the beginning of ceftazidime short infusion
C-reactive protein, leukocytes and hepatic enzymes levels at the beginning and the end of each IV antibiotic course

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Hubert, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (15):
- France (15):
  - CHU Grenoble, Grenoble
  - Centre hospitalier Dr Schaffner, Lens
  - Hopital Albert Calmette, Lille
  - Hopital Jeanne de Flandre, Lille
  - Hopital Sainte Marguerite, Marseille
  - Assistance Publique des hopitaux de paris, Hopital Trousseau, Paris
  - Assistance Publique des Hopitaux de Paris, Hopital Cochin, Paris
  - Assistance Publique des Hopitaux de Paris, Hopital Necker, Paris
  - Assistance Publique des Hopitaux de Paris, Hopital Robert Debré, Paris
  - Hopital Sud, Rennes
  - Centre Héliomarin, Roscoff
  - Hopital Hautepierre, Strasbourg
  - Hopital Foch, Suresnes
  - Hopital Larrey, Toulouse
  - Hopital de Brabois, Vandœuvre-lès-Nancy